CLINICAL TRIAL: NCT01962090
Title: A Comparison of Two Thoracic Manipulation Techniques to Improve Neck Pain in Dentistry Students: a Randomized Controlled Trial.
Brief Title: Comparison of Two Thoracic Manipulation Techniques to Improve Neck Pain in Dentistry Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A.T. Still University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000350
Record Dates: First submitted 2013-10-09; First posted 2013-10-14 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Neck Pain
Keywords: Neck Pain; Thoracic spine thrust manipulation; Osteopathic Manipulation; Dentistry; Range of Motion
MeSH Terms: conditions — Neck Pain | interventions — Sitting Position; Supine Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thoracic Spine Thrust in Seated Position (Experimental): Thoracic spine thrust manipulation will be applied two times at each of two treatment sessions while the participant is in a seated position.
  Interventions: Other: Thoracic Spine Thrust in Seated Position
- Thoracic Spine Thrust in Supine Position (Experimental): Thoracic spine thrust manipulation will be applied two times at each of two treatment sessions while the participant is in the supine position.
  Interventions: Other: Thoracic Spine Thrust in Supine Position

INTERVENTIONS:
Other: Thoracic Spine Thrust in Seated Position — The thoracic spine manipulation used here is a manipulation technique that involves positioning the patient so that a small amplitude quick stretch can be applied to the least mobile area of the thoracic spine as identified by the licensed physical therapist during spinal segmental mobility testing.
  Arms: Thoracic Spine Thrust in Seated Position
Other: Thoracic Spine Thrust in Supine Position — The thoracic spine manipulation used here is a manipulation technique that involves positioning the patient so that a small amplitude quick stretch can be applied to the least mobile area of the thoracic spine as identified by the licensed physical therapist during spinal segmental mobility testing.
  Arms: Thoracic Spine Thrust in Supine Position

SUMMARY:
This study is designed to compare the short term effects of two different thoracic spine thrust manipulation techniques on neck range of motion, pain, and self-reported disability in a sample of dental students experiencing neck pain.

The hypothesis of the study is that there will be a difference between the two thoracic spine thrust manipulation techniques for short term effects on neck range of motion, pain, and self-reported disability in a sample of dental students experiencing neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Current student at the Arizona School of Dentistry and Oral Health (ASDOH) at A. T. Still University
* Primary complaint of neck pain with or without symptoms that spread down into one arm
* Overall rating of neck pain intensity is at least 3/10; the overall rating is the overall average of the participant's rating of current, least, and worst pain experienced over the previous 24 hours on separate numeric pain rating scales where 0 corresponds to "no pain" and 10 corresponds to "worst pain possible".
* Neck Disability Index (NDI) score > 10 points (measure of self-reported disability with a 0 to 50 point scale where higher scores indicate higher levels of disability.
* Proficient in speaking and reading English to complete outcome questionnaires

Exclusion Criteria:

* Neck pain related to a motor vehicle accident or other trauma within the previous 6 weeks
* Neck pain that spreads down into both arms
* Low back pain or thoracic origin of pain
* Nerve root involvement; defined as the presence of two or more neurological findings (e.g. decreased strength, diminished deep tendon reflex, or decreased sensation) at the same nerve root level
* Diagnosis of cervical spine stenosis (narrowing of the central canal that contains the spinal cord)
* History of spinal tumors, spinal infection, cervical spine fracture, or previous neck surgery
* Pending legal action related to current episode of neck pain
* Contraindications to thoracic spine thrust manipulation

  1. serious pathologies or conditions (tumor, fracture, metabolic diseases, rheumatoid arthritis, osteoporosis, history of prolonged steroid use)
  2. hyperreflexia
  3. unsteadiness during gait
  4. Nystagmus
  5. Loss of visual acuity
  6. Impaired sensation of the face
  7. Altered taste
  8. The presence of pathological reflexes
  9. pregnancy or considering pregnancy

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2013-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in Neck Pain Intensity | Collected at baseline assessment during initial visit before 1st treatment, one week later before 2nd treatment, and one week later at follow-up appointment - total of 2- 3 weeks anticipated
  Each participant's neck pain intensity will be assessed by use of the Numeric Pain Rating Scale (NPRS of 0-10)
Change in Neck Range of Motion (ROM) | Collected at baseline assessment during initial visit before 1st treatment, one week later before 2nd treatment, and one week later at follow-up appointment - total of 2- 3 weeks anticipated
  Neck range of motion will be measured by a licensed Physical Therapist
Change in Neck Disability Index (NDI) | Collected at baseline assessment during initial visit before 1st treatment, one week later before 2nd treatment, and one week later at follow-up appointment - total of 2- 3 weeks anticipated
  The Neck Disability Index (NDI) is a self-reported measure of disability consisting of a 0-50 point scale where higher scores indicate higher levels of disability
Change in Shortened version of the Disabilities of the Arm, Shoulder, and Hand (QuickDASH) questionnaire (QuickDASH) | Collected at baseline assessment during initial visit before 1st treatment, one week later before 2nd treatment, and one week later at follow-up appointment - total of 2- 3 weeks anticipated
  The shortened version of the Disabilities of the Arm, Shoulder, and Hand (Quick DASH) questionnaire is a self-report measure of function that can assess how neck pain may be impacting daily activities that require use of the upper limb

CONTACTS AND LOCATIONS:
Overall Officials: John Heick, PT, DPT, Principal Investigator — A.T. Still University
Locations (1):
- A. T. Still University, Mesa, Arizona, United States